CLINICAL TRIAL: NCT00000170
Title: Amblyopia Treatment Study: Occlusion Versus Pharmacologic Therapy for Moderate Amblyopia
Brief Title: Occlusion Versus Pharmacologic Therapy for Moderate Amblyopia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEI-73; 2U10EY011751 (NIH); 5U10EY011751 (NIH)
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Amblyopia
Keywords: Amblyopia; patching; atropine
MeSH Terms: conditions — Amblyopia | interventions — Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patching (Active Comparator)
  Interventions: Device: Eye Patch
- Atropine (Active Comparator): Atropine
  Interventions: Drug: Atropine

INTERVENTIONS:
Drug: Atropine — Atropine
  Arms: Atropine
Device: Eye Patch — Patching
  Arms: Patching

SUMMARY:
* To determine whether the success rate with drug treatment (atropine) of amblyopia due to strabismus or anisometropia in patients less than 7 years old is equivalent to the success rate with occlusion (patching) therapy
* To develop more precise estimates of the success rates of amblyopia treatment
* To identify factors that may be associated with successful treatment of amblyopia
* To collect data on the course of treated amblyopia to provide more precise estimates of treatment effects than are now available

Extended Follow up of Study Patients

* Primary: To determine the long-term visual acuity outcome at age 10 years and at age 15 years in patients diagnosed with amblyopia before age 7 years.
* Secondary: To determine whether the long-term visual acuity outcome at age 10 years and at age 15 years differs between patients who received patching followed by best clinical care and patients who received atropine followed by best clinical care

DETAILED DESCRIPTION:
Amblyopia, or lazy eye, is the most common cause of visual impairment in children and often persists in adulthood. It is reported to be the leading cause of vision loss in one eye in the 20-70 year old age group, with a prevalence of 1-4 percent in various studies, indicating that both improved means of detection and treatment are needed.

Most of the available data on the natural history of amblyopia and success rates of its treatment with either patching or drug therapy are retrospective and uncontrolled. Despite the common occurrence of amblyopia, there is little quality data on treatment of this condition. Thus, there is much to be learned about the course of treated amblyopia, to provide more precise estimates of success rates and to identify factors that may be associated with successful and unsuccessful treatment.

Amblyopia, when diagnosed in children, is usually treated with occlusion (patching) of the sound eye. Occlusion therapy is subject to problems of compliance, due to the child's dislike of wearing a patch for visual, skin irritation, and social/psychological reasons. There is evidence that compliance may be one of, if not, the most important determinant of success of amblyopia therapy.

An alternative treatment, drug therapy with a cycloplegic drug (atropine) that dilates the pupils and blurs the image seen by the sound eye, has been known for almost a century. This method has been widely used for the management of occlusion treatment failures and for maintenance therapy. However, it has seen little use as a primary treatment for amblyopia. Clinical experience has found that it has a high acceptability to patients and parents, and hence high compliance. In addition to its acceptability, pharmacologic therapy has the known advantage over occlusion of providing a wider visual field with both eyes, which may have safety and other functional implications. There is also clinical and laboratory evidence suggesting that drug therapy may maintain and improve the ability to see with both eyes (binocularity).

Available data suggest that the success rate with drug therapy is as good as, if not better than, the success rate with occlusion therapy for mild to moderate degrees of amblyopia. If this is true, for many children with amblyopia, drug therapy may be the preferred initial therapy since it appears to be more readily accepted by the children and parents. Despite data to support the use of drug therapy as a primary therapy for amblyopia, it has gained only limited use among pediatric ophthalmologists. A definitive study comparing the outcomes from occlusion therapy and drug therapy is justified in order to determine if new practice guidelines for treatment of amblyopia are needed.

Regardless of whether the trial determines that one therapeutic approach is better than the other, the data that are collected will provide valuable information about the course of amblyopia treatment that is not presently available. The study also is expected to provide data that will help to determine whether factors such as age, refractive status, cause of amblyopia, or fixation pattern should be considered in determining which procedure is best for a given patient.

Extended Follow-up of Study Patients

The extended follow up study consists of annual visits prior to age 10, followed by a visit at age 10 years and a visit at age 15 years. There is no amblyopia treatment that is required during the extended follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 7 years old or younger with amblyopia due to strabismus or anisometropia
* Visual acuity in the amblyopic eye must be between 20/40 and 20/100
* Visual acuity in the sound eye or 20/40 or better
* At least 3 lines of acuity difference between the two eyes

Exclusion Criteria:

* More than two months of amblyopia therapy in the past two years
* Myopia (more than -0.50 D)

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 419 (Actual)
Dates: Start 1999-04; Primary Completion 2001-11 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Visual acuity in the amblyopic eye | 6 months

SECONDARY OUTCOMES:
Visual acuity in the amblyopic eye | 24 months
Extended Follow-up: (Primary) To determine the long-term visual acuity outcome at age 10 years and at age 15 years in patients diagnosed with amblyopia before age 7 years | age 10 years and age 15 years
Extended Follow-up: To determine whether the long-term visual acuity outcome at age 10 yrs and age 15 yrs differs between patients who received patching followed by best clinical care and patients who received atropine followed by best clinical care | age 10 years and age 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael X. Repka, M.D., Study Chair — Wilmer Eye Institute
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States

REFERENCES:
- [Background] Pediatric Eye Disease Investigator Group.. A randomized trial of atropine vs. patching for treatment of moderate amblyopia in children. Arch Ophthalmol. 2002 Mar;120(3):268-78. doi: 10.1001/archopht.120.3.268. PMID 11879129
- [Background] Pediatric Eye Disease Investigator Group. The clinical profile of moderate amblyopia in children younger than 7 years. Arch Ophthalmol. 2002 Mar;120(3):281-7. PMID 11879130
- [Background] Cole SR, Beck RW, Moke PS, Celano MP, Drews CD, Repka MX, Holmes JM, Birch EE, Kraker RT, Kip KE; Pediatric Eye Disease Investigator Group. The Amblyopia Treatment Index. J AAPOS. 2001 Aug;5(4):250-4. doi: 10.1067/mpa.2001.117097. PMID 11507585
- [Background] Holmes JM, Beck RW, Repka MX, Leske DA, Kraker RT, Blair RC, Moke PS, Birch EE, Saunders RA, Hertle RW, Quinn GE, Simons KA, Miller JM; Pediatric Eye Disease Investigator Group. The amblyopia treatment study visual acuity testing protocol. Arch Ophthalmol. 2001 Sep;119(9):1345-53. doi: 10.1001/archopht.119.9.1345. PMID 11545641
- [Background] Pediatric Eye Disease Investigator Group. A comparison of atropine and patching treatments for moderate amblyopia by patient age, cause of amblyopia, depth of amblyopia, and other factors. Ophthalmology. 2003 Aug;110(8):1632-7; discussion 1637-8. doi: 10.1016/S0161-6420(03)00500-1. PMID 12917184
- [Background] Pediatric Eye Disease Investigator Group. The course of moderate amblyopia treated with atropine in children: experience of the amblyopia treatment study. Am J Ophthalmol. 2003 Oct;136(4):630-9. doi: 10.1016/s0002-9394(03)00458-6. PMID 14516802
- [Background] Pediatric Eye Disease Investigator Group. The course of moderate amblyopia treated with patching in children: experience of the amblyopia treatment study. Am J Ophthalmol. 2003 Oct;136(4):620-9. doi: 10.1016/s0002-9394(03)00392-1. PMID 14516801
- [Background] Holmes JM, Beck RW, Kraker RT, Cole SR, Repka MX, Birch EE, Felius J, Christiansen SP, Coats DK, Kulp MT; Pediatric Eye Disease Investigator Group. Impact of patching and atropine treatment on the child and family in the amblyopia treatment study. Arch Ophthalmol. 2003 Nov;121(11):1625-32. doi: 10.1001/archopht.121.11.1625. PMID 14609923
- [Background] Repka MX, Wallace DK, Beck RW, Kraker RT, Birch EE, Cotter SA, Donahue S, Everett DF, Hertle RW, Holmes JM, Quinn GE, Scheiman MM, Weakley DR; Pediatric Eye Disease Investigator Group. Two-year follow-up of a 6-month randomized trial of atropine vs patching for treatment of moderate amblyopia in children. Arch Ophthalmol. 2005 Feb;123(2):149-57. doi: 10.1001/archopht.123.2.149. PMID 15710809
- [Background] Repka MX, Holmes JM, Melia BM, Beck RW, Gearinger MD, Tamkins SM, Wheeler DT; Pediatric Eye Disease Investigator Group. The effect of amblyopia therapy on ocular alignment. J AAPOS. 2005 Dec;9(6):542-5. doi: 10.1016/j.jaapos.2005.07.009. PMID 16414520
- [Background] Repka MX, Melia M, Eibschitz-Tsimhoni M, London R, Magoon E; Pediatric Eye Disease Investigator Group. The effect on refractive error of unilateral atropine as compared with patching for the treatment of amblyopia. J AAPOS. 2007 Jun;11(3):300-2. doi: 10.1016/j.jaapos.2006.09.017. PMID 17572346
- [Background] Pediatric Eye Disease Investigator Group; Repka MX, Kraker RT, Beck RW, Holmes JM, Cotter SA, Birch EE, Astle WF, Chandler DL, Felius J, Arnold RW, Tien DR, Glaser SR. A randomized trial of atropine vs patching for treatment of moderate amblyopia: follow-up at age 10 years. Arch Ophthalmol. 2008 Aug;126(8):1039-44. doi: 10.1001/archopht.126.8.1039. PMID 18695096
- [Background] Repka MX, Kraker RT, Beck RW, Cotter SA, Holmes JM, Arnold RW, Astle WF, Sala NA, Tien DR; Pediatric Eye Disease Investigator Group. Monocular oral reading performance after amblyopia treatment in children. Am J Ophthalmol. 2008 Dec;146(6):942-7. doi: 10.1016/j.ajo.2008.06.022. Epub 2008 Aug 16. PMID 18708179
- [Derived] Repka MX, Kraker RT, Holmes JM, Summers AI, Glaser SR, Barnhardt CN, Tien DR; Pediatric Eye Disease Investigator Group. Atropine vs patching for treatment of moderate amblyopia: follow-up at 15 years of age of a randomized clinical trial. JAMA Ophthalmol. 2014 Jul;132(7):799-805. doi: 10.1001/jamaophthalmol.2014.392. PMID 24789375
- [Derived] Kulp MT, Foster NC, Holmes JM, Kraker RT, Melia BM, Repka MX, Tien DR; Pediatric Eye Disease Investigator Group. Effect of ocular alignment on emmetropization in children <10 years with amblyopia. Am J Ophthalmol. 2012 Aug;154(2):297-302.e1. doi: 10.1016/j.ajo.2012.02.035. Epub 2012 May 23. PMID 22633344
- [Derived] Repka M, Simons K, Kraker R; Pediatric Eye Disease Investigator Group. Laterality of amblyopia. Am J Ophthalmol. 2010 Aug;150(2):270-4. doi: 10.1016/j.ajo.2010.01.040. Epub 2010 May 8. PMID 20451898